CLINICAL TRIAL: NCT05063734
Title: A Phase 2, Randomised, Multicentre Study to Assess the Dose Level of Multiple THR-687 Injections and to Evaluate the Efficacy and Safety of THR-687 Versus Aflibercept for the Treatment of Diabetic Macular Oedema (DME)
Brief Title: A Study to Evaluate THR-687 Treatment for Diabetic Macular Oedema.
Acronym: INTEGRAL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on data obtained in Part A, there was insufficient evidence of efficacy on the key outcome measures. As a result, the study was not advanced to Part B.
Sponsor: Oxurion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THR-687-002; 2020-000362-42 (EudraCT Number)
Record Dates: First submitted 2021-09-08; First posted 2021-10-01 (Actual); Results first posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus; Diabetic Retinopathy; Diabetic Macular Edema
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A, THR-687 1.2 mg (Experimental)
  Interventions: Drug: THR-687 dose level 1
- Part A, THR-687 2.0mg (Experimental)
  Interventions: Drug: THR-687 dose level 2
- Part B, treatment naïve subjects, THR-687 selected dose level (Experimental): Due to the discontinuation of the study after Part A, the dose level for Part B has not been selected
  Interventions: Drug: THR-687 selected dose level
- Part B, treatment naïve subjects, aflibercept 2.0mg (Active Comparator)
  Interventions: Drug: Aflibercept
- Part B, previously treated subjects, THR-687 selected dose level (Experimental): Due to the discontinuation of the study after Part A, the dose level for Part B has not been selected
  Interventions: Drug: THR-687 selected dose level
- Part B, previously treated subjects, aflibercept 2.0mg (Active Comparator)
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: THR-687 dose level 1 — 3 intravitreal injections of THR-687 dose level 1, 1 month apart
  Arms: Part A, THR-687 1.2 mg
Drug: THR-687 dose level 2 — 3 intravitreal injections of THR-687 dose level 2, 1 month apart
  Arms: Part A, THR-687 2.0mg
Drug: THR-687 selected dose level — 3 intravitreal injections of THR-687 selected dose level, 1 month apart, possibly followed by a 4th intravitreal injection with the same dose level of THR-687 at Month 3, or Month 4, or Month 5, if any of the PRN criteria are met.
  Arms: Part B, previously treated subjects, THR-687 selected dose level; Part B, treatment naïve subjects, THR-687 selected dose level
Drug: Aflibercept — 3 intravitreal injections of aflibercept, 1 month apart, possibly followed by a 4th intravitreal injection with aflibercept at Month 3, or Month 4, or Month 5, if any of the PRN criteria are met.
  Other Names: Eylea®
  Arms: Part B, previously treated subjects, aflibercept 2.0mg; Part B, treatment naïve subjects, aflibercept 2.0mg

SUMMARY:
This study is conducted to select the THR-687 dose level (Part A of the study) and to assess the efficacy and safety of the selected dose level compared to aflibercept (Part B of the study).

DETAILED DESCRIPTION:
In Part A, approximately 12 subjects are planned to be randomized (1:1 allocation) to THR-687 1.2mg and THR-687 2.0mg.

In Part B, in the cohort of Treatment Naïve subjects are planned to be randomized (2:1 allocation) to THR-687 selected dose level from Part A and Aflibercept 2.0mg.

In Part B, in the cohort of Previously Treated subjects are planned to be randomized (1:1 allocation) to THR-687 selected dose level from Part A and Aflibercept 2.0mg.

All subjects in the study will receive study treatment in one selected study eye only.

ELIGIBILITY:
The subjects in this study will be subjects with central-involved DME (CI-DME). Both treatment-naïve and previously treated subjects will be included.

Inclusion Criteria:

* Written informed consent obtained from the subject prior to screening procedures
* Male or female aged 18 years or older at the time of signing the informed consent
* Type 1 or type 2 diabetes
* BCVA ETDRS letter score ≥ 39 in the study eye
* CI-DME with CST of ≥ 300µm in men (or equivalent in women), measured from RPE to ILM inclusively, on SD-OCT, in the study eye
* BCVA ETDRS letter score ≥ 34 in the fellow eye

Exclusion Criteria:

* Macular edema due to causes other than DME in the study eye
* Concurrent disease in the study eye, other than DME, that could require medical or surgical intervention during the study period or could confound interpretation of the results
* Any condition in the study eye that could confound the ability to detect the efficacy of the investigational medicinal product
* Previous confounding medications / interventions, or their planned administration during the study
* Presence of iris neovascularisation in the study eye
* Uncontrolled glaucoma in the study eye
* Previously received THR-687 or any other experimental therapy for DME, in either eye
* Any active or suspected ocular or periocular infection, or active intraocular inflammation, in either eye
* Untreated Diabetes
* Glycated haemoglobin A (HbA1c) > 12%
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Department, Study Director — Oxurion
Locations (25):
- United States (18):
  - Salehi Retina Institute Inc., Huntington Beach, California
  - California Eye Specialists Medical Group, Inc., Pasadena, California
  - Retinal Consultants Medical Group, Sacramento, California
  - Retina Consultants of Southern Colorado, P.C., Colorado Springs, Colorado
  - Retina Associates, Ltd, Elmhurst, Illinois
  - University Retina and macula Associates, PC, Oak Forest, Illinois
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Sierra Eye Associates, Reno, Nevada
  - Retina Vitreous Surgeons of Central New York, PC, Liverpool, New York
  - Tulsa Retina Consultants, Tulsa, Oklahoma
  - Eye Care Specialists, Kingston, Pennsylvania
  - Tennessee Retina, PC, Nashville, Tennessee
  - Austin Research Center of Retina, Austin, Texas
  - Retina Consultants of Texas, Katy, Texas
  - Valley Retina Institute, P.A., McAllen, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina Center of Texas, Southlake, Texas
  - Strategic Clinical Research Group, Willow Park, Texas
- Estonia (2):
  - Eye Clinic Dr Krista Turman, Tallinn
  - Silmalaser OU, Tallinn
- Hungary (2):
  - Ganglion Medical Center, Pécs
  - Szegedi Tudományegyetem, Szeged
- Latvia (2):
  - Pauls Stradins Clinical University Hospital, Riga
  - Riga East Clinical University Hospital, Riga
- Vilnius University Hospital Santaros klinikos, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A, THR-687 1.2mg; Part A, THR-687 2.0mg: THR-687: 3 intravitreal injections of THR-687, 1 month apart
Period: Overall Study
Arm/Group | Part A, THR-687 1.2mg | Part A, THR-687 2.0mg
Started | 7 | 9
Completed | 6 | 9
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A, THR-687 1.2mg | Part A, THR-687 2.0mg | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (13.61) | 59.0 (9.55) | 62.6 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 3 | 6 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in BCVA ETDRS Letter Score, at Month 3, in Treatment-naïve Subjects in Part B of the Study
Time Frame: At Month 3
Population: Part B of the study was not initiated due to insufficient evidence of efficacy based on the data obtained in Part A
Groups:
- Part B, Treatment naïve Subjects, THR-687 Selected Dose Level: 3 intravitreal injections of THR-687 selected dose level, 1 month apart, possibly followed by a 4th intravitreal injection with the same dose level of THR-687 at Month 3, or Month 4, or Month 5, if any of the PRN criteria are met
- Part B, Treatment naïve Subjects, Aflibercept: 3 intravitreal injections of aflibercept, 1 month apart, possibly followed by a 4th intravitreal injection with aflibercept at Month 3, or Month 4, or Month 5, if any of the PRN criteria are met
Arm/Group | Part B, Treatment naïve Subjects, THR-687 Selected Dose Level | Part B, Treatment naïve Subjects, Aflibercept
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Weighted Average of the Change From Baseline in BCVA ETDRS Letter Score From Day 8 Through Month 3 Using the Trapezoidal Rule (AUC), in Treatment-naïve Subjects in Part B of the Study
Time Frame: at Month 3
Population: Part B of the study was not initiated due to insufficient evidence of efficacy based on the data obtained in Part A
Arm/Group | Part B, Treatment naïve Subjects, THR-687 Selected Dose Level | Part B, Treatment naïve Subjects, Aflibercept
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in BCVA ETDRS Letter Score, by Study Visit, in Treatment-naïve Subjects in Part B of the Study
Time Frame: Up to Month 8
Population: Part B of the study was not initiated due to insufficient evidence of efficacy based on the data obtained in Part A
Arm/Group | Part B, Treatment naïve Subjects, THR-687 Selected Dose Level | Part B, Treatment naïve Subjects, Aflibercept
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in Central Subfield Thickness (CST), Based on Spectral Domain Optical Coherence Tomography (SD-OCT), as Assessed by the Central Reading Center (CRC), by Study Visit, in Treatment-naïve Subjects in Part B of the Study
Time Frame: Up to Month 8
Population: Part B of the study was not initiated due to insufficient evidence of efficacy based on the data obtained in Part A
Arm/Group | Part B, Treatment naïve Subjects, THR-687 Selected Dose Level | Part B, Treatment naïve Subjects, Aflibercept
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Incidence of Ocular and Non-ocular Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Adverse Events will be reported from the date of Informed Consent until End of the Study visit (up to Month 6 in Part A and up to Month 8 in Part B) or at the early study discontinuation visit and will be coded using MedDRA. Adverse Events will be summarized by System Organ Class and Primary Term. Incidence by subject represents at least one occurrence of the Primary Term with an onset on or after the date of the first study treatment. If a subject has multiple occurrences of an adverse event (P-term), the subject is presented only once in the respective subject count.
Time Frame: Up to End of Study (Part A up to Month 6 and Part B up to Month 8)
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, THR-687 1.2mg | Part A, THR-687 2.0mg
Number analyzed (Participants) | 7 | 9
Participants | 4 | 6

ADVERSE EVENTS:
Time Frame: Up to End of Study (up to Month 6 for Part A and up to Month 8 for Part B)
Description: All Adverse Events were collected from the time the subject provided consent to participate in the study until the end of the study (last study visit) for the subject.
Arm/Group | Part A, THR-687 1.2mg | Part A, THR-687 2.0mg
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/9
Other Adverse Events (participants affected / at risk) | 4/7 | 6/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, THR-687 1.2mg (N=7) | Part A, THR-687 2.0mg (N=9)
Cataract Subcapsular (Eye disorders) | 0 (0) | 1 (1)
Diabetic Retinal Oedema (Eye disorders) | 0 (0) | 1 (1)
Optic Disc Haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Posterior Capsule Opacification (Eye disorders) | 0 (0) | 1 (1)
Retinal Thickening (Eye disorders) | 0 (0) | 3 (3)
Visual Acuity Reduced (Eye disorders) | 1 (1) | 3 (3)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Intraocular Pressure Increased (Investigations) | 0 (0) | 1 (2)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
Genital Disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
Based on data obtained in Part A, there was insufficient evidence of efficacy on the key outcome measures. As a result, the study was not advanced to Part B

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/34/NCT05063734/Prot_SAP_000.pdf